CLINICAL TRIAL: NCT05635773
Title: The Role of a Visual Alexa Enabled Visual Device in Aiding Performance in Emergency Front-of-Neck Access (eFONA-A) Within a Simulated 'Can't Intubate Can't Oxygenate' Scenario
Brief Title: Use of Alexa as a Cognitive Aid for Emergency Front Of Neck Access (FONA)
Acronym: FONA-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: IRAS 266480
Record Dates: First submitted 2022-04-19; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-04

CONDITIONS: Intubation; Difficult or Failed

STUDY DESIGN:
Intervention Model Description: Randomisation will be carried out using a randomization table made at www.randomizer.org to even/odd allocation numbers corresponding to 'Alexa first' vs 'No Alexa first' group with equal allocation between each arm. The randomisation sequence will be known only to the investigators issuing the initial grouping to the candidate, and allocations will be concealed from the video recording assessors and the statistical analysis team.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Assessors marking the recorded performances will be blinded as to which group the candidate had been allocated to in the first instance. The statistical analysis team will also be blinded to the allocation sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eFONA No Alexa (Active Comparator): Arm randomised to performing the procedure without Alexa cognitive aid first
  Interventions: Device: Use of Alexa Visual Cognitive aid
- eFONA Alexa (Experimental): Arm randomised to performing the procedure using Alexa cognitive aid first
  Interventions: Device: Use of Alexa Visual Cognitive aid

INTERVENTIONS:
Device: Use of Alexa Visual Cognitive aid — The intervention is the use of of a cognitive aid to determine the efficacy of the aid in completing the steps correctly.

SUMMARY:
The aim of the study is to investigate whether a voice activated cognitive aid can improve performance in a simulated emergency front-of-neck access scenario. This skill is ideally practiced on an annual basis by anaesthetists in training, with a variety of usually low-fidelity simulation used.

The addition of the Alexa cognitive aid is a novel step with the aim of improving adherence to the recommended steps required to successfully complete the procedure. One arm of this study will be introduced to the Alexa checklist in advance of performing the procedure prior to crossover, whereas the second arm will not (subject to standard anaesthetic training).

ELIGIBILITY:
Inclusion Criteria:

* CT1 to Consultant level Anaesthetists, who have completed the Initial Assessment of Competencies (IAC)

Exclusion Criteria:

* Anaesthetists without the above criteria, refusal

Min Age: 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
The number of critical steps missed. | 6 months
  What critical steps were missed

SECONDARY OUTCOMES:
All critical steps completed | 6 months
  What critical steps were completed
Hypoxic time (interval between SpO2 first <94% to recover >=94% - explicitly timed gradual decrease in saturations) | 6 months
  What was the hypoxic time
A measure of participant workload (e.g. NASA-TLX) as perceived and completed by the participant after each arm. | 6 months
  Workload time versus perceived time per participant
A measure of team working (e.g. ANTS score) for each individual procedure | 6 months
  Actual measure per participant per procedure
A measure of participant's subjective experience (e.g. qualitative analysis of participant feedback on the device) | 6 months
  Feedback from each participant about the device

CONTACTS AND LOCATIONS:
Overall Officials: Craig Johnstone, MBChB, Principal Investigator — Guy's & St Thomas' NHS Trust
Locations (1):
- Guy's & St Thomas' NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided